CLINICAL TRIAL: NCT04962880
Title: Prevalence of Homologous Recombination Repair (HRR) Gene Mutations in Patients With Metastatic Castration-resistant Prostate Cancer in Latin America: PROSPECT Study.
Brief Title: HRR Prevalence in LatAm PROSPECT Study
Acronym: PROSPECT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D081LR00003
Record Dates: First submitted 2021-06-17; First posted 2021-07-15 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Castration-resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Archived FFPE tumor blocks (tissue sample) from eligible participants will be requested from the local pathology laboratory and used for HRR mutation testing. A blood sample will be taken from each participant enrolled in the study independently of the FFPE availability. Blood sample must be available for testing under the algorithm of this protocol. After checking FFPE tissue availability Pathologist will perform an assessment in order to check sample quality. If pathology assessment of FFPE sample accomplishes sample quality requirements tissue will be cut in 5um slices and 15 to 20 slides will be provided to reference laboratory.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determine the prevalence of homologous recombination repair (HRR) gene mutations in participants with mCRPC in Latin America (LatAm) between February 2021 and January 2022.

DETAILED DESCRIPTION:
Background/Rationale: Prostate cancer(PC)is the second most frequent cancer diagnosis made in men and the fifth leading cause of death worldwide(1). Variations in the incidence rates world wide reflect differences in multiple epidemiological variables depending on the different regions. It is known that in Central America is the leading cause of cancer death in men. For South America, it is the second cause of cancer death and the third in North America(2). Estimations from 2012 from Brazil reported over 60,000 new cases. While in 2017 the United States (US) reported more than 160,000 new cases, represent in gone in five diagnosis of cancer in men (3-5).

The incidence of castration-resistant prostate cancer (CRPC)has been reported in several studies in various regions of the world, but unfortunately in Latin America data are incomplete. A comprehensive systematic review including 71,179 patients observed for up to 12 years, indicated that 10.0-20.0% of PC patients developed CRPC within approximately five years of follow-up. Over 84.0% of them had metastases present at the time of CRPC diagnosis, and 33.0% of those without metastases at diagnosis developed them within two years (3,4). Currently, patients with metastatic CRPC (mCRPC) have an overall survival rate between 9 and 13 months and is associated with bone metastases and poor quality of life (3.7). The negative prognosis of mCRPC may be associated in part with few and limited therapeutic options. In the past decade, there have been few new treatment options for this group of patients becoming an unmet need, but the development of targeted therapies and the application of PCD-damaged DNA repair mutation detection (DDR) tests allow patient classification and offer them important treatment options, particularly in advanced stages of the disease where current options are limited (8,9).

Objectives and Hypotheses Primary Objective: Determine the prevalence of homologous recombination repair (HRR) gene mutations in participants with mCRPC in Latin America(LatAm) between February 2021 and January 2022.

Exploratory objectives

1. Describe the demographic and clinical characteristics of the mCRPC participants with HRR gene mutations in LatAm between February 2021 and January 2022.
2. Describe the association between demographic and clinical characteristics, and the prevalence of HRR gene mutations in participants with mCRPC per LatAm country between February 2021 and January 2022.

No hypothesis will be considered for the study.

Methods:

Study design: A cross-sectional, non-interventional, multicenter study to determine the prevalence of HRR gene mutations in participants with metastatic castration-resistant prostate cancer in LatAm. The study will be performed in reference centers for the attention of mCRPC patients in LatAm countries (Argentina, Brazil, Colombia, Costa Rica, Mexico, Panama and Peru). The study will select participants with mCRPC diagnosed between February 2021 and January 2022.

During screening visit, consecutive eligible participants who have been diagnosed with mCRPC will be invited to participate, and after consent, their demographic in formation and history of cancer data will be collected. Archived FFPE tumor blocks (tissue sample)from eligible participants will be requested from the local pathology laboratory and used for HRR mutation testing. A blood sample will be taken from each participant enrolled in the study independently of the FFPE availability-. Although blood sample must be available for testing under the algorithm of this protocol, not all blood samples will be processed and/ or analyzed. After checking FFPE tissue availability Pathologist will perform an assessment in order to check sample quality. If pathology assessment of FFPE sample accomplishes sample quality requirements tissue will be cut in 5um slices and 15 to 20 slides will be provided to reference laboratory.

After NGS sequencing and complete analyses are performed for each sample, reporting will be performed signed from Laboratory main investigator. Reporting will be delivered to Participant ́s Center and Physician will report the results to each participant.

Participants' medical records will be reviewed for data relevant to mCRPC diagnosis, including basic demographic information, medical history, and treatment history. Approximately 390 patients will be enrolled in this study. It is anticipated that participants will be enrolled at eight sites in multiple countries, including Argentina, Brazil, Colombia, CostaRica, Mexico, Panama and Peru(Panama and Costa Rica, and Colombia and Peru are considered as clusters).The maximum duration of the study is expected to be 12months.

Data Source(s):To perform HRR mutation testing, archival FFPE biopsy tissue samples from primary or metastatic tumor will be used. HRR genes according to provider ́s protocol. FFPE slides and blood samples will be analysed using New Generation Sequencing (NGS) at one central analytics laboratory (reference laboratory) in each country. Each reference laboratory will perform HRR mutation testing and report mutation status of each of the genes included in the test according to the procedure established by the HRR mutation testing manufacturer. Variants classification will be performed according ACMG guidelines. All demographic informationandhistoryofcancerdata(includingprevioustreatments)fromparticipantswill be collected in retrospective manner using patient medical records. Data will be entered in the electronic forms. The principal investigator will be responsible for ensuring that all required data are collected and entered into the electronic forms.

Study Population :Study population will be the diagnosed castration resistant metastatic prostate cancer patients in the selected countries from February 2021 and January 2022..It is estimated that approximately 390 patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged≥18
2. Pathological mCRPC cases confirmed by histopathological report.
3. Evidence of a previous methastatic primary PC
4. Availability to provide medical history data(demographic information and history of cancer).
5. Availability to provide blood and/or tissue sample in case it is available
6. Participants who are able to sign the informed consent form(ICF).

Exclusion Criteria:

1. Diagnosis of any severe acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of the study results
2. Inability of participant to provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males will be consider for this study.
Study Population: Study population will be the diagnosed castration-resistant metastatic prostate cancer patients in the selected countries
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | Q1 2021 - Q1 2022
  To know the prevalence and type of Homologous Recombinational Repair (HRR) mutations identified in Formalin-fixed paraffin-embedded (FFPE) tissue or blood samples in patients diagnosed with metastatic castration-resistant prostate cancer (mCRPC) in the selected participants countries in LatAm.
  A molecular test formulary would be completed when tissue sample is analyzed
  * Preservation time (years)
  * Origin of the FFPE (organ)
  * HRR mutation status (32 mutations would be analyzed and each of them would have as an answer "positive"/"negative"/"VUS")
  A molecular test formulary would be completed when blood sample is analyzed
  * Date of extraction (date)
  * HRR mutation status (32 mutations would be analyzed and each of them would have as an answer "positive"/"negative"/"VUS")

OTHER OUTCOMES:
Exploratory Outcomes | Q1 2021 - Q1 2022
  Demographic and clinical characteristics of mCRPC participants with HRR mutations in LatAm.
  * Date of birth (day/month/year)
  * Race (white, black, asian, afroamerican, hispanic, mestizo)
  * Country of origin
  * Family history of cancer (type, year of diagnosis, degree of kinship)
  * mCRPC diagnosis (year)
  * Metastasis location (several options)
  * Other medical condition (type, start year, end year)
  * ECOG evaluation (0 to 4)
  * Performance Status
  * Treatment (several options)
  * Sample collected (tissue /blood)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Garbaos, MD, Principal Investigator — Fundación Estudios Clinicos; Martin Angel, MD, Principal Investigator — INSTITUTO ALEXANDER FLEMING; Ray Manneh Kopp, MD, Principal Investigator — Sociedad de Oncología y Hematología del Cesar S.A.S.; Jorge A Chaves Porras, MD, Principal Investigator — Instituto de Investigaciones en Ciencias Médicas (ICIMED); Alejandro Crismatt, MD, Principal Investigator — Centro Hemato Oncológico Panamá (CHOP); Silvia Neciosup, MD, Principal Investigator — Centro de Investigación Oncosalud - RCI N° 166; Miguel A Álvarez Avitia, MD, Principal Investigator — Instituto Nacional de Cancerología (INCAN); Arturo Delgado Herrera, MD, Principal Investigator — Centro Médico Nacional Siglo XXI (CMNSXXI); Pedro H Isaacsson Velho, MD, Principal Investigator — Centro de Pesquisa Hospital Moinhos de Vento
Locations (11):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Rosario
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Research Site, Bogotá, Colombia
- Research Site, San José, Costa Rica
- Mexico (2):
  - Research Site, Mexico City, Mexico DF
  - Research Site, Mexico City
- Research Site, Panama City, Panama
- Research Site, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081LR00003&attachmentIdentifier=74911adf-d526-4b42-b1b4-7f174b700da6&fileName=D081LR00003_CSR_Synopsis.pdf&versionIdentifier=